CLINICAL TRIAL: NCT05096221
Title: A Phase 3 Multinational, Randomized, Double-Blind, Placebo-Controlled Systemic Gene Delivery Study to Evaluate the Safety and Efficacy of SRP-9001 in Subjects With Duchenne Muscular Dystrophy (EMBARK)
Brief Title: A Gene Transfer Therapy Study to Evaluate the Safety and Efficacy of Delandistrogene Moxeparvovec (SRP-9001) in Participants With Duchenne Muscular Dystrophy (DMD)
Acronym: EMBARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRP-9001-301; 2019-003374-91 (EudraCT Number)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Muscular Dystrophies; Duchenne Muscular Dystrophy; DMD; North Star Ambulatory Assessment (NSAA); Ambulatory; Pediatric; Gene-Delivery
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delandistrogene Moxeparvovec followed by Placebo (Experimental): Participants will receive single intravenous (IV) infusion of delandistrogene moxeparvovec on Day 1. Then, participants will receive a single IV infusion of matching placebo at Year 2.
  Interventions: Genetic: delandistrogene moxeparvovec; Genetic: placebo
- Placebo followed by Delandistrogene Moxeparvovec (Placebo Comparator): Participants will receive matching placebo IV infusion on Day 1. Then, participants will have the opportunity to receive a single IV infusion of delandistrogene moxeparvovec at Year 2.
  Interventions: Genetic: delandistrogene moxeparvovec; Genetic: placebo

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec.
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS
Genetic: placebo — Single IV infusion of matching placebo.

SUMMARY:
The study will evaluate the safety and efficacy of gene transfer therapy in boys with DMD. It is a randomized, double-blind, placebo-controlled study. The participants who are randomized to the placebo arm will have an opportunity for treatment with gene transfer therapy at the beginning of the second year.

ELIGIBILITY:
Inclusion Criteria:

* Is ambulatory and from 4 to under 8 years of age at time of randomization.
* Definitive diagnosis of DMD based on documented clinical findings and prior genetic testing.
* Ability to cooperate with motor assessment testing.
* Stable daily dose of oral corticosteroids for at least 12 weeks prior to Screening, and the dose is expected to remain constant throughout the study (except for modifications to accommodate changes in weight).
* rAAVrh74 antibody titers are not elevated as per protocol-specified requirements.
* A pathogenic frameshift mutation or premature stop codon contained between exons 18 and 79 (inclusive), with the exception of mutation fully contained within exon 45.

Exclusion Criteria:

* Exposure to gene therapy, investigational medication, or any treatment designed to increase dystrophin expression within protocol specified time limits.
* Abnormality in protocol-specified diagnostic evaluations or laboratory tests.
* Presence of any other clinically significant illness, medical condition, or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risk for gene transfer.

Other inclusion or exclusion criteria could apply.

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (42):
- United States (23):
  - Arkansas Children's, Little Rock, Arkansas
  - UC San Diego Altman Clinical and Translational Research Institute, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University of St. Louis, St Louis, Missouri
  - Columbia University/NYPH, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Lenox Baker Children's Hospital, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Wisconsin, Milwaukee, Wisconsin
- University Hospital Ghent, Ghent, Belgium
- Germany (3):
  - LMU - Klinikum der Universitaet Muenchen - Kinderklinik und, Bayern
  - Universitätsklinikum Essen - Klinik für Kinderheilkunde I, Essen
  - University Hospital Hamburg- Eppendorf, Hamburg
- Hong Kong Children's Hospital, Kowloon, Hong Kong
- Italy (3):
  - IRCCS Istituto G.Gaslini, U.O., Genoa
  - UOC Neurologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - UOC Neuropsichiatria Infantile, Area Salute del Bambino, Fondazione Policlinico Universitario A. Gamelli IRCCS, Roma
- Japan (4):
  - Kobe University Hospital, Kobe
  - National Center for Child Health and Development, Tokyo
  - Tokyo Women's Medical University Hospital - Pediatrics, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
- Spain (2):
  - Hospital Universitari i Politécnico La Fe, Valencia, Comunidad Valencia
  - Hospital Sant Joan de Déu, Barcelona
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - Oxford University Hospitals NHS Foundation Trust, Headington, Oxford
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - The Newcastle Upon Tyne NHS Hospital NHS Foundation Trust, Royal Victoria Infirmary, Newcastle upon Tyne

REFERENCES:
- [Result] Mendell JR, Muntoni F, McDonald CM, Mercuri EM, Ciafaloni E, Komaki H, Leon-Astudillo C, Nascimento A, Proud C, Schara-Schmidt U, Veerapandiyan A, Zaidman CM, Guridi M, Murphy AP, Reid C, Wandel C, Asher DR, Darton E, Mason S, Potter RA, Singh T, Zhang W, Fontoura P, Elkins JS, Rodino-Klapac LR. AAV gene therapy for Duchenne muscular dystrophy: the EMBARK phase 3 randomized trial. Nat Med. 2025 Jan;31(1):332-341. doi: 10.1038/s41591-024-03304-z. Epub 2024 Oct 9. PMID 39385046
- [Derived] Mendell JR, Muntoni F, McDonald CM, Mercuri EM, Ciafaloni E, Komaki H, Leon-Astudillo C, Nascimento A, Proud C, Schara-Schmidt U, Veerapandiyan A, Zaidman CM, Furgerson M, Ding K, Singh P, Potter R, Asher DR, Murphy AP, Reid C, Hooper G, Torre CO, Manfrini M, Rodino-Klapac LR. Two-Year Outcomes Following Delandistrogene Moxeparvovec Treatment in Ambulatory Patients with Duchenne Muscular Dystrophy: Phase 3 EMBARK Trial. Neurol Ther. 2026 Jan 10. doi: 10.1007/s40120-025-00879-8. Online ahead of print. PMID 41518520
- [Derived] Audhya I, Nacson AB, Gooch K, Basnyat B, Slota C, Martin S, Murphy A, Lansdall CJ, Ciobanu T, Nascimento A, Veerapandiyan A. Caregiver-reported Patient Experiences with Duchenne Muscular Dystrophy: Qualitative In-trial Interviews 1 Year After Delandistrogene Moxeparvovec in the Pivotal EMBARK Trial. Neurol Ther. 2025 Nov 3. doi: 10.1007/s40120-025-00842-7. Online ahead of print. PMID 41182527
- [Derived] Vandenborne K, Walter GA, Straub V, Willcocks RJ, Forbes SC, Mercuri EM, Muntoni F, Ding K, Ennamuri S, Reid C, Murphy AP, Manfrini M, Mendell JR, Elkins JS, Rodino-Klapac LR. Quantitative Muscle Magnetic Resonance Outcomes in Patients With Duchenne Muscular Dystrophy: An Exploratory Analysis From the EMBARK Randomized Clinical Trial. JAMA Neurol. 2025 Jul 1;82(7):734-744. doi: 10.1001/jamaneurol.2025.0992. PMID 40354061
- [Derived] McDonald CM, Elkins JS, Dharmarajan S, Gooch K, Ciobanu T, Lansdall CJ, Murphy AP, McDougall F, Mercuri EM, Audhya I; EMBARK Study Group. Caregiver Global Impression Observations from EMBARK: A Phase 3 Study Evaluating Delandistrogene Moxeparvovec in Ambulatory Patients with Duchenne Muscular Dystrophy. Neurol Ther. 2025 Feb;14(1):211-225. doi: 10.1007/s40120-024-00685-8. Epub 2024 Nov 26. PMID 39589719
- See also: SRP-9001-301 Plain Language Study Summary — https://www.sarepta.com/sites/sarepta-corporate/files/2025-06/SRP-9001-301_English_PLSS.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 126 participants were enrolled in the study. 1 of the 126 participants was enrolled via a country-specific protocol addendum. Data are presented below for the 125 participants enrolled via the global protocol.
Groups:
- Delandistrogene Moxeparvovec Followed by Placebo: Participants received a single intravenous (IV) infusion of delandistrogene moxeparvovec on Day 1 of Part 1. Then, participants received a single IV infusion of matching placebo on Day 1 in Part 2.
- Placebo Followed by Delandistrogene Moxeparvovec: Participants received a single IV infusion of matching placebo on Day 1 of Part 1. Then, participants received a single IV infusion of delandistrogene moxeparvovec on Day 1 in Part 2.
Period: Part 1
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Started | 63 | 62
Received at Least 1 Dose of Study Drug in Part 1 | 63 | 62
Completed | 63 | 62
Not Completed | 0 | 0
Period: Part 2
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Started | 63 | 60 (Two participants who completed Part 1 discontinued prior to Part 2.)
Received at Least 1 Dose of Study Drug in Part 2 | 62 | 60
Completed | 63 | 59
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Measured in the Modified Intent-to-Treat (mITT) Population, which included all randomized participants who received study treatment, with treatment group designated according to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.98 (1.06) | 6.08 (1.05) | 6.03 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 63 | 62 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 8 | 23
  Not Hispanic or Latino | 47 | 53 | 100
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 11 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black of African American | 0 | 2 | 2
  White | 49 | 46 | 95
  More than One Race | 1 | 0 | 1
  Other or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in North Star Ambulatory Assessment (NSAA) Total Score at Week 52
Description: The NSAA is a healthcare provider administered scale that rates performance of various motor abilities in ambulant children with Duchenne Muscular Dystrophy and is used to monitor disease progression and treatment effects. During assessment, participants are asked to perform 17 different functional activities that are graded as: 2 - "Normal" - no obvious modification of activity; 1 - Modified method but achieves goal independent of assistance; 0 - Unable to achieve independently. The NSAA total score is defined as the sum of all 17 items, ranging from 0 (worst) to 34 (best). The response vector consists of the change from baseline in NSAA total score at the post-baseline visit. The model includes the covariates of treatment group, visit, treatment group by visit interaction, age group, baseline NSAA total score, and baseline NSAA total score by visit interaction. All covariates are fixed effects in this analysis. An increase in score indicates an improvement in motor function.
Time Frame: Baseline, Week 52 (Part 1)
Population: Measured in the Modified Intent-to-Treat (mITT) Population, which included all randomized participants who received study treatment, with treatment group designated according to randomization. Here, "Number of Participants Analyzed"= number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 63 | 61
scores on a scale | 2.57 (0.39) | 1.92 (0.39)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.2441, Mixed model of repeated measures; Least squares mean change difference = 0.65, 95% CI 2-sided [-0.45 to 1.74], Standard Error of Mean 0.55

2. Secondary Outcome: Part 1: Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression at Week 12 as Measured by Western Blot Adjusted by Muscle Content
Description: Quantity of delandistrogene moxeparvovec dystrophin protein levels (in muscle biopsy samples) were determined by Western blot at Part 1, Week 12. For this endpoint, 2 blocks of tissues were analyzed by Western blot, each with 2 technical replicates to determine the delandistrogene moxeparvovec dystrophin protein level (percent control). The block average value from 2 technical replicates was computed. The overall average was calculated as the mean of the block average values. The overall average values were used for the analysis. Dystrophin protein was measured and then adjusted based on the percentage of muscle content in the biopsy sample. An increase in protein expression indicates production of the delandistrogene moxeparvovec dystrophin protein.
Time Frame: Week 12
Population: Measured in the mITT Population, which included all randomized participants who received study treatment, with treatment group designated according to randomization. Here, "Number of Participants Analyzed"= number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent control
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 17 | 14
Percent control | 34.29 (41.04) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Other; p < 0.0001, Re-randomization test

3. Secondary Outcome: Part 1: Change From Baseline in Time to Rise From the Floor at Week 52
Description: The time to rise from the floor test quantifies the time required for the participant to stand in an upright position with arms by sides, starting from the supine position with arms by sides. Data are presented for the change from baseline to Week 52 in the time taken (in seconds) to rise from the floor.
Time Frame: Baseline, Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 63 | 61
Seconds | -0.27 (0.15) | 0.37 (0.15)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.0025, Mixed model of repeated measures; Least squares mean change difference = -0.64, 95% CI 2-sided [-1.06 to -0.23], Standard Error of Mean 0.21

4. Secondary Outcome: Part 1: Change From Baseline in Time to Complete 10 Meter Walk/Run (10MWR) at Week 52
Description: The timed 10MWR quantifies the time required for the participant to run or walk 10 meters (on a straight walkway) from a standing position. Data are presented for change from baseline to Week 52 in the time (in seconds) taken to complete the 10MWR.
Time Frame: Baseline, Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 63 | 61
Seconds | -0.34 (0.10) | 0.08 (0.10)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.0048, Mixed model of repeated measures; Least squares mean change difference = -0.42, 95% CI 2-sided [-0.71 to -0.13], Standard Error of Mean 0.15

5. Secondary Outcome: Part 1: Change From Baseline in Time to Complete 100 Meter Walk/Run (100MWR) at Week 52
Description: The timed 100MWR quantifies the time required for the participant to run or walk 100 meters (on a straight walkway) from a standing position. Data are presented for change from baseline to Week 52 in the time (in seconds) taken to complete the 100MWR.
Time Frame: Baseline, Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 59 | 57
Seconds | -6.57 (1.76) | -3.28 (1.80)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.1942, Mixed model of repeated measures; Least squares mean change difference = -3.29, 95% CI 2-sided [-8.28 to 1.70], Standard Error of Mean 2.52

6. Secondary Outcome: Part 1: Change From Baseline in the Timed Stair Ascend 4 Steps Test at Week 52
Description: The timed stair ascend 4 steps test quantifies the time required for the participant to ascend 4 standard steps (each step was 6 inches in height). Data presented is the change from baseline to Week 52 in the time (in seconds) to ascend 4 steps.
Time Frame: Baseline, Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 62 | 60
Seconds | -0.44 (0.12) | -0.08 (0.13)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.0412, Mixed model of repeated measures; Least squares mean change difference = -0.36, 95% CI 2-sided [-0.71 to -0.01], Standard Error of Mean 0.18

7. Secondary Outcome: Part 1: Change From Baseline in Stride Velocity 95th Centile (SV95C) at Week 52
Description: Each participant was provided with wearable devices to collect data on stride velocity. Participants wore a device on each ankle. SV95C data was derived based on stride velocity. Data are presented for change from baseline to Week 52 in SV95C.
Time Frame: Baseline, Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: meters (m)/second (s)
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 57 | 61
meters (m)/second (s) | 0.06 (0.03) | -0.03 (0.03)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.0402, Mixed model of repeated measures; Least squares mean change difference = 0.10, 95% CI 2-sided [0.00 to 0.19], Standard Error of Mean 0.05

8. Secondary Outcome: Part 1: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Score in Mobility to Week 52
Description: PROMIS is a family of instruments developed and validated to assess health-related quality of life, including mobility. Mobility function scores ranged from 1 (worst mobility function) to 5 (best mobility function), where higher scores indicate a better clinical outcome.
Time Frame: Baseline, Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 57 | 59
Scores on a scale | 0.05 (0.05) | -0.01 (0.05)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.4272, Mixed model of repeated measures; Least squares mean change difference = 0.05, 95% CI 2-sided [-0.08 to 0.19], Standard Error of Mean 0.07

9. Secondary Outcome: Part 1: Change From Baseline in PROMIS Score in Upper Extremity Function to Week 52
Description: PROMIS is a family of instruments developed and validated to assess health-related quality of life, including upper extremity function. Upper extremity function scores ranged from 1 (not able to do so [worst upper extremity function]) to 5 (no trouble [best upper extremity function]), where higher scores indicate a better clinical outcome.
Time Frame: Baseline, Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 57 | 58
scores on a scale | 0.19 (0.07) | 0.23 (0.07)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.7324, Mixed model of repeated measures; Least squares mean change difference = -0.04, 95% CI 2-sided [-0.24 to 0.17], Standard Error of Mean 0.10

10. Secondary Outcome: Part 1: Number of Skills Gained or Improved at Week 52 as Measured by the NSAA
Description: The NSAA is a clinician-administered scale that rates performance on various functional activities. As measured by the NSAA, data was collected for the number of skills gained (the average item score was 0 at Baseline and > 0 at Part 1 Week 52) or improved (the average item score at Baseline was > 0 but less than the average item score at Part 1 Week 52). As pre-specified, data are presented for the combined number of skills gained or improved at Week 52.
Time Frame: Week 52 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of skills
Arm/Group | Delandistrogene Moxeparvovec Followed by Placebo | Placebo Followed by Delandistrogene Moxeparvovec
Number analyzed (Participants) | 63 | 61
number of skills | 4.18 (0.31) | 3.99 (0.31)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Followed by Placebo vs Placebo Followed by Delandistrogene Moxeparvovec; Test type: Superiority; p = 0.6554, Mixed model of repeated measures; Least squares mean change difference = 0.19, 95% CI 2-sided [-0.67 to 1.06], Standard Error of Mean 0.44

11. Secondary Outcome: Parts 1 and 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as an adverse event (AE) that emerged during treatment, having been absent pre-treatment, or worsened relative to the pretreatment state. SAEs were defined as any adverse event that resulted in death, was life threatening, required or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or was an important medical event. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 104 weeks
Population: Measured in the Safety Population in Part 1, which included all participants who received study treatment, with treatment group designated according to the treatment they received. Measured in the SRP-treated population in Part 2, which included all participants who received investigational study treatment (delandistrogene moxeparvovec) in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Delandistrogene Moxeparvovec in Part 1 Followed by Placebo in Part 2: Participants received a single intravenous (IV) infusion of delandistrogene moxeparvovec on Day 1 of Part 1. Then, participants received a single IV infusion of matching placebo on Day 1 in Part 2.
- Part 1: Placebo in Part 1 Followed by Delandistrogene Moxeparvovec in Part 2; Part 2: Placebo in Part 1 Followed by Delandistrogene Moxeparvovec in Part 2: Participants received a single IV infusion of matching placebo on Day 1 of Part 1. Then, participants received a single IV infusion of delandistrogene moxeparvovec on Day 1 in Part 2.
- Part 2: Delandistrogene Moxeparvovec in Part 1 Followed by Placebo in Part 2: Participants received a single IV infusion of delandistrogene moxeparvovec on Day 1 of Part 1. Then, participants received a single IV infusion of matching placebo on Day 1 in Part 2.
Arm/Group | Part 1: Delandistrogene Moxeparvovec in Part 1 Followed by Placebo in Part 2 | Part 1: Placebo in Part 1 Followed by Delandistrogene Moxeparvovec in Part 2 | Part 2: Delandistrogene Moxeparvovec in Part 1 Followed by Placebo in Part 2 | Part 2: Placebo in Part 1 Followed by Delandistrogene Moxeparvovec in Part 2
Number analyzed (Participants) | 63 | 62 | 63 | 60
Participants
  TEAEs | 62 | 57 | 53 | 56
  SAEs | 14 | 5 | 5 | 8

12. Secondary Outcome: Parts 1 and 2: Number of Participants With Adverse Events of Special Interest (AESI)
Description: AESIs were defined as adverse events (AEs) of special interest, based on pre-specified criteria and pertain to categories labeled hepatotoxicity, immune-mediated myositis, thrombotic microangiopathy (TMA), hypersensitivity, thrombocytopenia, rhabdomyolysis, and troponin I elevations. The data represent the number of participants who experienced an event within the specified AESI category as observed by the principal investigator (PI), after adjudication. Per prespecified analysis, AESI data were only collected based on the specified AESI categories. A Summary of all SAEs and nonserious AEs ("Other"), regardless of causality and regardless of the AESI category, is located in the "Reported Adverse Events" section.
Time Frame: Up to 104 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Delandistrogene Moxeparvovec in Part 1 Followed by Placebo in Part 2 | Part 1: Placebo in Part 1 Followed by Delandistrogene Moxeparvovec in Part 2 | Part 2: Delandistrogene Moxeparvovec in Part 1 Followed by Placebo in Part 2 | Part 2: Placebo in Part 1 Followed by Delandistrogene Moxeparvovec in Part 2
Number analyzed (Participants) | 63 | 62 | 63 | 60
Participants
  Hepatotoxicity | 12 | 0 | 0 | 14
  Immune-mediated Myositis | 0 | 0 | 0 | 0
  TMA | 0 | 0 | 0 | 0
  Hypersensitivity | 1 | 0 | 1 | 0
  Thrombocytopenia | 2 | 0 | 1 | 0
  Rhabdomyolysis | 1 | 1 | 0 | 0
  Troponin I elevations | 2 | 1 | 14 | 8

ADVERSE EVENTS:
Time Frame: Up to approximately 104 weeks
Description: Part 1: data are reported in the Safety Population, which included all participants who received study treatment, with treatment group designated according to the treatment they received. Part 2: data are reported in the SRP-treated population, which included all participants who received investigational study treatment (delandistrogene moxeparvovec) in the study.
Groups:
- Part 1: Delandistrogene Moxeparvovec: Participants received a single IV infusion of delandistrogene moxeparvovec on Day 1 of Part 1.
- Part 1: Placebo: Participants received a single IV infusion of matching placebo on Day 1 of Part 1.
- Part 2: Placebo: Participants who received delandistrogene moxeparvovec on Day 1 of Part 1 received a single IV infusion of matching placebo on Day 1 in Part 2.
- Part 2: Delandistrogene Moxeparvovec: Participants who received matching placebo on Day 1 in Paty 1 received a single IV infusion of delandistrogene moxeparvovec on Day 1 in Part 2.
Arm/Group | Part 1: Delandistrogene Moxeparvovec | Part 1: Placebo | Part 2: Placebo | Part 2: Delandistrogene Moxeparvovec
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/62 | 0/63 | 0/60
Serious Adverse Events (participants affected / at risk) | 14/63 | 5/62 | 5/63 | 8/60
Other Adverse Events (participants affected / at risk) | 62/63 | 57/62 | 52/63 | 55/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Delandistrogene Moxeparvovec (N=63) | Part 1: Placebo (N=62) | Part 2: Placebo (N=63) | Part 2: Delandistrogene Moxeparvovec (N=60)
COVID-19 (Infections and infestations) | 2 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Toxic shock syndrome streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 2
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Prescription drug used without a prescription (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Delandistrogene Moxeparvovec (N=63) | Part 1: Placebo (N=62) | Part 2: Placebo (N=63) | Part 2: Delandistrogene Moxeparvovec (N=60)
Vomiting (Gastrointestinal disorders) | 39 | 11 | 9 | 43
Nausea (Gastrointestinal disorders) | 24 | 8 | 5 | 23
Abdominal pain upper (Gastrointestinal disorders) | 10 | 9 | 1 | 11
Diarrhoea (Gastrointestinal disorders) | 6 | 13 | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 0 | 8
Constipation (Gastrointestinal disorders) | 5 | 5 | 4 | 6
COVID-19 (Infections and infestations) | 15 | 10 | 6 | 6
Upper respiratory tract infection (Infections and infestations) | 13 | 17 | 10 | 13
Influenza (Infections and infestations) | 9 | 3 | 2 | 5
Nasopharyngitis (Infections and infestations) | 9 | 12 | 4 | 5
Ear infection (Infections and infestations) | 6 | 6 | 2 | 4
Enterobiasis (Infections and infestations) | 5 | 0 | 5 | 1
Viral infection (Infections and infestations) | 5 | 5 | 5 | 2
Gastroenteritis viral (Infections and infestations) | 4 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 2 | 4 | 1 | 1
Pyrexia (General disorders) | 19 | 14 | 5 | 12
Fatigue (General disorders) | 9 | 6 | 1 | 10
Glutamate dehydrogenase increased (Investigations) | 18 | 2 | 1 | 12
Gamma-glutamyltransferase increased (Investigations) | 5 | 0 | 2 | 12
Blood creatine phosphokinase increased (Investigations) | 1 | 4 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 20 | 3 | 1 | 15
Irritability (Psychiatric disorders) | 9 | 4 | 2 | 3
Aggression (Psychiatric disorders) | 1 | 4 | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 7 | 9 | 5 | 5
Fall (Injury, poisoning and procedural complications) | 5 | 7 | 5 | 6
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 4 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 19 | 12 | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 7 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 12 | 8 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 2 | 8
Headache (Nervous system disorders) | 8 | 8 | 9 | 10
Cushingoid (Endocrine disorders) | 4 | 4 | 0 | 3
Gastroenteritis (Infections and infestations) | 0 | 2 | 4 | 2
Troponin I increased (Investigations) | 2 | 2 | 6 | 5
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 6
Joint injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3
Attention deficit hyperactivity disorder (Psychiatric disorders) | 4 | 1 | 3 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 4
Proteinuria (Renal and urinary disorders) | 1 | 0 | 4 | 2
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 4
Seasonal allergy (Immune system disorders) | 3 | 2 | 4 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT05096221/Prot_SAP_001.pdf